CLINICAL TRIAL: NCT02752334
Title: The Effect on Outcome of Adding Magnesium Sulphate to Bupivacaine in the Ultrasound-guided Supraclavicular Brachial Plexus Block Anesthesia
Brief Title: Magnesium Sulphate in the Ultrasound-guided Supraclavicular Brachial Plexus Block
Acronym: Mg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Magrabi Eye & Ear Hospital (Other)
Responsible Party: Principal Investigator, Ashraf M Ghali, proffesor of anesthesia and ICU, Magrabi Eye & Ear Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MEEC-IRB-2016-1
Record Dates: First submitted 2016-03-03; First posted 2016-04-26 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group Bupivacaine (No Intervention): patients will receive 23 mL of Bupivacaine HCL 0.5% (Marcaine, 5 mg per mL; Hospira, USA) in addition to 2 mL normal saline using Ultrasound-guided Supraclavicular Brachial Plexus Block
- group Bupivacaine Magnesium (Active Comparator): patients will receive 23 mL of Bupivacaine HCL 0.5% in addition to 2 mL (100 mg) Magnesium Sulphate (Magnesium Sulphate 50 %, 500 mg per mL; Hospira, USA) diluted with normal saline. using Ultrasound-guided Supraclavicular Brachial Plexus Block
  Interventions: Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Magnesium Sulphate — Magnesium has antinociceptive effects in animal and human models, principally related to blocking the N-methyl-D-aspartate (NMDA) receptors and regulation of calcium influx into cells.
  Other Names: Bupivacaine HCL 0.5%
  Arms: group Bupivacaine Magnesium

SUMMARY:
This study evaluated the motor and sensory block duration and the postoperative analgesic effects of adding Magnesium Sulphate to bupivacaine in the ultrasound-guided supraclavicular brachial plexus block Anesthesia. Motor and sensory block duration were considered as a primary endpoint.

DETAILED DESCRIPTION:
The supraclavicular approach to the brachial plexus provides more consistent and effective regional anesthesia to the upper extremity than other approaches to brachial plexus blockade. However, the fear of pneumothorax is often cited by anesthetists as a reason to avoid this approach. With increasing affirmation on patient safety and better patient outcomes, ultrasound guided regional anesthesia (UGRA) is becoming more widely popular. Ultrasound provides clinicians with a real time image suitable for visualizing anatomical structures, needle placement, and local anesthetic spread. Ultrasound-guidance to supraclavicular brachial plexus block has shown to increase success rates, reduce the volume of local anesthetic (LA) used and has the potential to minimize the risk of complications.

Although there are many treatment choices for postoperative pain, a gold standard has not been established. Prolonging the duration of peripheral nerve blocks using long-acting Local Anesthesia or perineural catheters can be used. However, perineural catheters are more time-consuming, costly, has possible higher complication rates (e.g. Infection), and needs more postoperative care.

Several adjuvants such as fentanyl, alpha-2 adrenergic agonists (clonidine or dexmedetomidine), tramadol, and magnesium have been used to extend the duration of peripheral nerve blocks. 5-7 Magnesium has antinociceptive effects in animal and human models, principally related to blocking the N-methyl-D-aspartate (NMDA) receptors and regulation of calcium influx into cells. Calcium influx leads to a sequence of central sensitization such as windup phenomenon and long term potentiation which are crucial mechanisms that determine the duration and intensity of post-operative pain. Magnesium prevents central sensitization triggered by peripheral nociceptive stimulation in response to painful stimuli.

The investigators designed this study to evaluate the effect of adding magnesium sulphate to bupivacaine in the ultrasound-guided supraclavicular brachial plexus block anesthesia. The sensory and motor block durations were evaluated as primary endpoints and the postoperative analgesic effects as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. - ASA physical status I to II,
2. - Patients listed for elective forearm or hand surgery using supraclavicular brachial plexus block anesthesia

Exclusion Criteria:

1 - evidence of severe cardiovascular, renal, or hepatic diseases, preexisting neurological or psychiatric illnesses.

2- patients have allergy to the study drugs. 3 - patients who have any contraindications to brachial plexus block anesthesia.

4- pregnant or lactating women, or 5- if the BMI was > 35 kg/m2.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The sensory block duration (the time interval between the end of local anesthetic administration and restoration of normal sensation) were evaluated as primary endpoint | 12 hours
  extended

SECONDARY OUTCOMES:
the postoperative analgesic effects (the time interval between the end of local anesthetic administration and the first analgesia given) as a secondary endpoint. | 12 hours
  improved

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M Ghali, Phd, Study Chair — Magrabi Eye & Ear Hospital
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
yes

REFERENCES:
- [Background] Tran DQ, Russo G, Munoz L, Zaouter C, Finlayson RJ. A prospective, randomized comparison between ultrasound-guided supraclavicular, infraclavicular, and axillary brachial plexus blocks. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):366-71. doi: 10.1097/AAP.0b013e3181ac7d18. PMID 19574871